CLINICAL TRIAL: NCT02943070
Title: NxThera Benign Prostatic Hyperplasia Rezum System Pilot Study
Brief Title: Rezum I Pilot Study for Benign Prostatic Hyperplasia
Acronym: Rezum Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1189-001
Record Dates: First submitted 2012-10-16; First posted 2016-10-24 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Prostatic Hyperplasia; Benign Prostatic Hyperplasia; Adenoma, Prostatic; Prostatic Adenoma; Prostatic Hyperplasia, Benign; Prostatic Hypertrophy; Prostatic Hypertrophy, Benign; Rezum
Keywords: Rezum; Water Vapor Ablation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rezum Treatment (Experimental): Patients received the Rezum transurethral needle ablation procedure to treat benign prostatic hyperplasia.
  Interventions: Device: Rezum System

INTERVENTIONS:
Device: Rezum System — The Rezūm System treats patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death. The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
  Other Names: Rezum Procedure; Rezum; Water Vapor Ablation; Rezum Delivery Device; Rezum Generator

SUMMARY:
Evaluate the safety and efficacy of the Rezum System for the treatment of BPH

DETAILED DESCRIPTION:
Prospective, non-randomized clinical trial of subjects with benign prostatic hyperplasia. The objective of the study are to 1) determine the safety and efficacy of the BPH Rezum System and assess its effect on urinary symptoms secondary to benign prostatic hyperplasia (BPH), and 2) further document the safety and post-operative effects of the Rezum System in the treatment of obstructive BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects > 45 years of age who have symptomatic / obstructive symptoms secondary to BPH requiring invasive intervention.
2. IPSS score of ≥ 15.
3. Qmax: Peak flow rate ≤ 15 ml/sec.
4. Post-void residual (PVR) < 300 ml.
5. Prostate transverse diameter > 30 mm.
6. Prostate volume between 20 to 120 gm.
7. Voided volume ≥ 125 mL
8. Subject able to complete the study protocol in the opinion of the investigator.
9. Life expectancy of at least one year.

Exclusion Criteria:

1. History of any illness or surgery that may confound the results of the study or have risk to subject.
2. Presence of a penile implant.
3. Any prior minimally invasive intervention (e.g. TUNA, Balloon, Microwave) or surgical intervention for the symptoms of BPH.
4. Currently enrolled or has been enrolled in another trial in the past 30 days.
5. Confirmed or suspected malignancy of prostate or bladder
6. Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease.
7. Previous pelvic irradiation or radical pelvic surgery.
8. Documented active urinary tract infection by culture or bacterial prostatitis within last year documented by culture (UTI is defined as >100,000 colonies per ml urine from midstream clean catch or catherization specimen)
9. Neurogenic bladder or sphincter abnormalities.
10. Urethral strictures, bladder neck contracture or muscle spasms.
11. Bleeding disorder or is currently on coumadin. (Note that use of anti-platelet medication is not an exclusion criteria.)
12. Subjects interested in maintaining fertility.
13. Use of concomitant medications to include the following:

    1. Use of, antihistamines, and antispasmodics within 1 week of treatment unless there is documented evidence stable dosing for last 6 months (no dose changes).
    2. Use of alpha blockers, androgens, or gonadotropin-releasing hormonal analogs within 2 weeks of treatment.
    3. Use of 5-alpha reductase inhibitor within the last 6 months
    4. Use of antidepressants, anticholinergics, anticonvulsants, and beta blockers unless there is documented evidence of stable dosing
14. Subject is unable or unwilling to go through the "washout" period prior to treatment.
15. Subject has chronic urinary retention.
16. Post-void residual volume > 300 ml.
17. Significant urge incontinence.
18. Poor detrusor muscle function.
19. Neurological disorders which might affect bladder or sphincter function.
20. Urinary sphincter abnormalities.
21. Bladder stones.
22. Evidence of bacterial prostatitis or symptoms of epididymitis
23. Renal impairment or serum creatinine > 2.0 mg/dl
24. In the physician's opinion, subject cannot tolerate a cystoscopy procedure well.
25. Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with all the required follow-up requirements.
26. Any cognitive disorder that interferes with or precludes direct and accurate communication with the study investigator regarding the study.
27. Peripheral arterial disease with intermittent claudication or Leriches Syndrome (i.e., claudication of the buttocks or perineum).
28. Biopsy of prostate within 30 days of procedure.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Hagelin, Study Director — Program Manager, Clinical Affairs, Boston Scientific
Locations (3):
- University Hospital, Brno, Czechia
- Clinica Canela, La Romana, Dominican Republic
- Urologcentrum, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, international, multicenter, non-randomized study recruited subjects who met inclusion/exclusion criteria and consented to participate. Subjects on BPH medication underwent a washout period prior to treatment. Subjects who successfully completed the washout period and still met the inclusion/exclusion criteria were enrolled in the study. Subjects were considered officially enrolled only if treatment with the NxThera Rezūm System was attempted.
Groups:
- Rezum Treatment: Subjects received the Rezum transurethral needle ablation procedure to treat benign prostatic hyperplasia.
  Rezum System: The Rezūm System treats patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death. The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
Period: Overall Study
Arm/Group | Rezum Treatment
Started | 50
Completed | 7
Not Completed | 43
Not completed — Physician Decision | 1
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4
Not completed — Retreatment or TURP | 13
Not completed — Subjects exited after their 48 month visit per the Sponsor's decision to close the study. | 18

BASELINE CHARACTERISTICS:
Population: Consecutive subjects who met inclusion/exclusion criteria and consented to participate were enrolled and treated with the NxThera Rezūm System.
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Black or African Origin | 2
  Ethnicity: Caucasian | 45
  Ethnicity: Hispanic or Latino | 3
Region of Enrollment [Number; unit: participants]
  Sweden | 27
  Czechia | 18
  Dominican Republic | 5

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS) Change From Baseline
Description: International Prostate Symptom Score (IPSS) scores were recorded at Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, then annually to 5 years. The mean change (improvement) in IPSS was calculated. IPSS scores range from 0 (no symptoms) to 35 (severe symptoms). Improvement in symptoms is shown by a reduction in score.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Mean change (improvement) in score was calculated for the number of subjects providing data at each follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  IPSS Change at 1 Week: number analyzed (Participants) | 49
  IPSS Change at 1 Week | -0.4 (7.8)
  IPSS Change at 1 Month: number analyzed (Participants) | 49
  IPSS Change at 1 Month | -5.0 (8.3)
  IPSS Change at 3 Months: number analyzed (Participants) | 48
  IPSS Change at 3 Months | -13.1 (7.2)
  IPSS Change at 6 Months: number analyzed (Participants) | 48
  IPSS Change at 6 Months | -12.6 (7.9)
  IPSS Change at 12 Months: number analyzed (Participants) | 45
  IPSS Change at 12 Months | -12.2 (7.7)
  IPSS Change at 24 Months: number analyzed (Participants) | 35
  IPSS Change at 24 Months | -11.7 (8.4)
  IPSS Change at 36 Months: number analyzed (Participants) | 27
  IPSS Change at 36 Months | -9.4 (9.0)
  IPSS Change at 48 Months: number analyzed (Participants) | 26
  IPSS Change at 48 Months | -9.6 (7.5)
  IPSS Change at 60 Months: number analyzed (Participants) | 7
  IPSS Change at 60 Months | -8.4 (6.7)

2. Primary Outcome: Major Complications
Description: Safety assessed by the frequency of systemic and local serious device related complications and the occurrence of unanticipated device-related adverse effects during treatment and at follow-up, up to 30 days. Due to the nature of the device, any device-related AEs are expected to present themselves during the immediate peri-procedure period (30 days post procedure).
  The device related complications that will be compared for this safety endpoint are:
  1. Severe Urinary Retention (Retention ≥ 24 hours)
  2. Fistula between rectum and urethra
  3. Perforation of the rectum or GI tract
  4. New incidences of retrograde ejaculation
Time Frame: 3 months
Population: Incidence of device-related complications pre-specified under this safety endpoint assessed through 3 months post-implant.
Measure: Number; unit: clinically relevant complications
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
clinically relevant complications
  Severe urinary retention (retention >=24 hours | 1
  Fistula between rectum and urethra | 0
  Perforation of the Rectum or GI Tract | 0
  New incidences of retrograde ejaculation | 0

3. Secondary Outcome: Proportion of Responders - Responders With a ≥ 30% International Prostate Symptom Score (IPSS) Improvement
Description: The proportion of study subjects who were responders were evaluated. A responder is defined as a subject with ≥ 30% improvement in BPH symptoms from baseline as measured by the IPSS.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Subjects with data at baseline and at the follow-up visit are included in the data summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Proportion of Responders with>=30% Improvement at 1 Week: number analyzed (Participants) | 49
  Proportion of Responders with>=30% Improvement at 1 Week | 12
  Proportion of Responders with>=30% Improvement at 1 Month: number analyzed (Participants) | 49
  Proportion of Responders with>=30% Improvement at 1 Month | 20
  Proportion of Responders with>=30% Improvement at 3 Months: number analyzed (Participants) | 48
  Proportion of Responders with>=30% Improvement at 3 Months | 39
  Proportion of Responders with>=30% Improvement at 6 Months: number analyzed (Participants) | 48
  Proportion of Responders with>=30% Improvement at 6 Months | 40
  Proportion of Responders with>=30% Improvement at 12 Months: number analyzed (Participants) | 45
  Proportion of Responders with>=30% Improvement at 12 Months | 36
  Proportion of Responders with>=30% Improvement at 24 Months: number analyzed (Participants) | 35
  Proportion of Responders with>=30% Improvement at 24 Months | 28
  Proportion of Responders with>=30% Improvement at 36 Months: number analyzed (Participants) | 27
  Proportion of Responders with>=30% Improvement at 36 Months | 19
  Proportion of Responders with>=30% Improvement at 48 Months: number analyzed (Participants) | 26
  Proportion of Responders with>=30% Improvement at 48 Months | 18
  Proportion of Responders with>=30% Improvement at 60 Months: number analyzed (Participants) | 7
  Proportion of Responders with>=30% Improvement at 60 Months | 4

4. Secondary Outcome: Proportion of Responders - Responders With a ≥ 50% International Prostate Symptom Score (IPSS) Improvement
Description: The proportion of study subjects who were responders were evaluated. For this measure a responder is defined as a subject with ≥ 50% improvement in BPH symptoms from baseline as measured by the IPSS.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Subjects with data at baseline and follow-up visits are included in the data summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Proportion of Responders with a ≥ 50% IPSS Improvement at 1 Week: number analyzed (Participants) | 49
  Proportion of Responders with a ≥ 50% IPSS Improvement at 1 Week | 3
  Proportion of Responders with a ≥ 50% IPSS Improvement at 1 Month: number analyzed (Participants) | 49
  Proportion of Responders with a ≥ 50% IPSS Improvement at 1 Month | 14
  Proportion of Responders with a ≥ 50% IPSS Improvement at 3 Months: number analyzed (Participants) | 48
  Proportion of Responders with a ≥ 50% IPSS Improvement at 3 Months | 35
  Proportion of Responders with a ≥ 50% IPSS Improvement at 6 Months: number analyzed (Participants) | 48
  Proportion of Responders with a ≥ 50% IPSS Improvement at 6 Months | 35
  Proportion of Responders with a ≥ 50% IPSS Improvement at 12 Months: number analyzed (Participants) | 45
  Proportion of Responders with a ≥ 50% IPSS Improvement at 12 Months | 30
  Proportion of Responders with a ≥ 50% IPSS Improvement at 24 Months: number analyzed (Participants) | 35
  Proportion of Responders with a ≥ 50% IPSS Improvement at 24 Months | 20
  Proportion of Responders with a ≥ 50% IPSS Improvement at 36 Months: number analyzed (Participants) | 27
  Proportion of Responders with a ≥ 50% IPSS Improvement at 36 Months | 15
  Proportion of Responders with a ≥ 50% IPSS Improvement at 48 Months: number analyzed (Participants) | 26
  Proportion of Responders with a ≥ 50% IPSS Improvement at 48 Months | 13
  Proportion of Responders with a ≥ 50% IPSS Improvement at 60 Months: number analyzed (Participants) | 7
  Proportion of Responders with a ≥ 50% IPSS Improvement at 60 Months | 2

5. Secondary Outcome: Proportion of Responders - Responders With Improvement ≥ 8 Points in IPSS
Description: Analysis will be provided for proportion of subjects with improvement ≥ 8 points from baseline at 1 week, 1 month, and 3 months, 6 months, 1 year, annually to 5 years
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 1 Week: number analyzed (Participants) | 49
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 1 Week | 9
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 1 Month: number analyzed (Participants) | 49
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 1 Month | 18
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 3 Months: number analyzed (Participants) | 48
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 3 Months | 37
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 6 Months: number analyzed (Participants) | 48
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 6 Months | 37
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 12 Months: number analyzed (Participants) | 45
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 12 Months | 33
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 24 Months: number analyzed (Participants) | 35
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 24 Months | 24
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 36 Months: number analyzed (Participants) | 27
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 36 Months | 17
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 48 Months: number analyzed (Participants) | 26
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 48 Months | 16
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 60 Months: number analyzed (Participants) | 7
  Proportion of Responders With Improvement ≥ 8 Points in IPSS at 60 Months | 4

6. Secondary Outcome: Uroflow Assessment - Change From Baseline in Peak Urinary Flow (Qmax)
Description: Peak urinary flow rate (Qmax) is the maximum urinary flow rate. It is calculated as milliliters (ml) of urine passed per second. Average results are based on age and sex. Typical uroflow rates ranges from 10 ml to 21 ml per second. An increase in mL/sec corresponds to improved urinary function.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Mean change in urinary flow rate was calculated for subjects with data at baseline and follow-up visit.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
mL/sec
  Change from baseline in peak urinary flow rate (Qmax) at 1 Week: number analyzed (Participants) | 47
  Change from baseline in peak urinary flow rate (Qmax) at 1 Week | -0.2 (4.3)
  Change from baseline in peak urinary flow rate (Qmax) at 1 Month: number analyzed (Participants) | 48
  Change from baseline in peak urinary flow rate (Qmax) at 1 Month | 1.9 (4.8)
  Change from baseline in peak urinary flow rate (Qmax) at 3 Months: number analyzed (Participants) | 47
  Change from baseline in peak urinary flow rate (Qmax) at 3 Months | 5.5 (6.6)
  Change from baseline in peak urinary flow rate (Qmax) at 6 Months: number analyzed (Participants) | 46
  Change from baseline in peak urinary flow rate (Qmax) at 6 Months | 5.2 (5.7)
  Change from baseline in peak urinary flow rate (Qmax) at 12 Months: number analyzed (Participants) | 45
  Change from baseline in peak urinary flow rate (Qmax) at 12 Months | 4.7 (7.0)
  Change from baseline in peak urinary flow rate (Qmax) at 24 Months: number analyzed (Participants) | 34
  Change from baseline in peak urinary flow rate (Qmax) at 24 Months | 4.1 (6.7)
  Change from baseline in peak urinary flow rate (Qmax) at 36 Months: number analyzed (Participants) | 26
  Change from baseline in peak urinary flow rate (Qmax) at 36 Months | 3.5 (6.2)
  Change from baseline in peak urinary flow rate (Qmax) at 48 months: number analyzed (Participants) | 9
  Change from baseline in peak urinary flow rate (Qmax) at 48 months | 3.0 (4.3)
  Change from baseline in peak urinary flow rate (Qmax) at 60 Months: number analyzed (Participants) | 6
  Change from baseline in peak urinary flow rate (Qmax) at 60 Months | 3.9 (4.3)

7. Secondary Outcome: Uroflow Assessment - Proportion of Subjects With Qmax Improvement of ≥ 30% From Baseline
Description: Peak urinary flow rate (Qmax) is the maximum urinary flow rate. It is calculated as milliliters (ml) of urine passed per second. This measure reports the number of subjects who experienced a ≥ 30% improvement from baseline at each follow-up interval.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Measure calculated for subjects with data at baseline and follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Qmax improvement of 30% or more over baseline at 1 Week: number analyzed (Participants) | 47
  Qmax improvement of 30% or more over baseline at 1 Week | 14
  Qmax improvement of 30% or more over baseline at 1 Month: number analyzed (Participants) | 48
  Qmax improvement of 30% or more over baseline at 1 Month | 21
  Qmax improvement of 30% or more over baseline at 3 Months: number analyzed (Participants) | 47
  Qmax improvement of 30% or more over baseline at 3 Months | 28
  Qmax improvement of 30% or more over baseline at 6 Months: number analyzed (Participants) | 46
  Qmax improvement of 30% or more over baseline at 6 Months | 32
  Qmax improvement of 30% or more over baseline at 12 Months: number analyzed (Participants) | 45
  Qmax improvement of 30% or more over baseline at 12 Months | 30
  Qmax improvement of 30% or more over baseline at 24 Months: number analyzed (Participants) | 34
  Qmax improvement of 30% or more over baseline at 24 Months | 20
  Qmax improvement of 30% or more over baseline at 36 Months: number analyzed (Participants) | 26
  Qmax improvement of 30% or more over baseline at 36 Months | 13
  Qmax improvement of 30% or more over baseline at 48 months: number analyzed (Participants) | 9
  Qmax improvement of 30% or more over baseline at 48 months | 4
  Qmax improvement of 30% or more over baseline at 60 Months: number analyzed (Participants) | 6
  Qmax improvement of 30% or more over baseline at 60 Months | 4

8. Secondary Outcome: Uroflow Assessment - Proportion of Subjects With Qmax Improvement of ≥ 3 ml/Sec
Description: Peak urinary flow rate (Qmax) is the maximum urinary flow rate. It is calculated as milliliters (ml) of urine passed per second. This measure reports the number of subjects who experienced a ≥3 mL/sec improvement from baseline at each follow-up interval.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Measure calculated for subjects with data at baseline and follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 1 Week: number analyzed (Participants) | 47
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 1 Week | 11
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 1 Month: number analyzed (Participants) | 48
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 1 Month | 19
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 3 Months: number analyzed (Participants) | 47
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 3 Months | 30
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 6 Months: number analyzed (Participants) | 46
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 6 Months | 30
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 12 Months: number analyzed (Participants) | 45
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 12 Months | 27
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 24 Months: number analyzed (Participants) | 34
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 24 Months | 18
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 36 Months: number analyzed (Participants) | 26
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 36 Months | 12
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 48 months: number analyzed (Participants) | 9
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 48 months | 3
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 60 Months: number analyzed (Participants) | 6
  Subjects with Qmax Improvement of ≥ 3 ml/sec at 60 Months | 3

9. Secondary Outcome: Uroflow Assessment - Change in Post Void Residual (PVR) by Follow up Interval
Description: Change in post void residual (PVR) urine volume in ml. Post void residual volume was measured by either ultrasound to measure the volume left in the bladder after urination, or by inserting a urinary catheter into the bladder after urination to drain and measure residual urine. Either measurement tool was allowed but the same measurement was to be used pre and post treatment.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Measure calculated for subjects with data at baseline and follow-up visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
ml
  Change from baseline in PVR at 1 Week: number analyzed (Participants) | 48
  Change from baseline in PVR at 1 Week | 48.8 (135.9)
  Change from baseline in PVR at 1 Month: number analyzed (Participants) | 48
  Change from baseline in PVR at 1 Month | -20.2 (94.7)
  Change from baseline in PVR at 3 Months: number analyzed (Participants) | 47
  Change from baseline in PVR at 3 Months | -30.5 (72.4)
  Change from baseline in PVR at 6 Months: number analyzed (Participants) | 46
  Change from baseline in PVR at 6 Months | -27.1 (81.6)
  Change from baseline in PVR at 12 Months: number analyzed (Participants) | 45
  Change from baseline in PVR at 12 Months | -22.8 (83.7)
  Change from baseline in PVR at 24 Months: number analyzed (Participants) | 34
  Change from baseline in PVR at 24 Months | -11.8 (102.2)
  Change from baseline in PVR at 36 Months: number analyzed (Participants) | 26
  Change from baseline in PVR at 36 Months | 11.9 (134.4)
  Change from baseline in PVR at 48 months: number analyzed (Participants) | 9
  Change from baseline in PVR at 48 months | -14.3 (54.5)
  Change from baseline in PVR at 60 Months: number analyzed (Participants) | 5
  Change from baseline in PVR at 60 Months | -12.6 (52.4)

10. Secondary Outcome: Change in Sexual Function - Erectile Function
Description: Change from baseline in sexual function was measured by the International Index of Erectile Function (IIEF) (Scoring on the IIEF ranges from 1 to 30. An increase in score indicates improvement from baseline)
Time Frame: 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Mean change in total score was calculated for subjects providing data at each follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  IEFF change from baseline at 1 Month: number analyzed (Participants) | 37
  IEFF change from baseline at 1 Month | -4.2 (20.7)
  IEFF change from baseline at 3 Months: number analyzed (Participants) | 40
  IEFF change from baseline at 3 Months | 3.3 (20.0)
  IEFF change from baseline at 6 Months: number analyzed (Participants) | 39
  IEFF change from baseline at 6 Months | 6.3 (17.6)
  IEFF change from baseline at 12 Months: number analyzed (Participants) | 39
  IEFF change from baseline at 12 Months | 5.8 (16.4)
  IEFF change from baseline at 24 Months: number analyzed (Participants) | 21
  IEFF change from baseline at 24 Months | 8.2 (14.8)
  IEFF change from baseline at 36 Months: number analyzed (Participants) | 15
  IEFF change from baseline at 36 Months | 10.7 (16.9)
  IEFF change from baseline at 48 Months: number analyzed (Participants) | 16
  IEFF change from baseline at 48 Months | 2.7 (27.4)
  IEFF change from baseline at 60 Months: number analyzed (Participants) | 4
  IEFF change from baseline at 60 Months | 12.5 (24.1)

11. Secondary Outcome: Change in Sexual Function - Retrograde Ejaculation
Description: Rate of Retrograde Ejaculation (when no fluid exits the penis during orgasm (e.g., dry orgasm)
Time Frame: 1 Week post procedure, 1 Month post procedure, 3 Months post procedure
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Incidence of retrograde ejaculation at 1 Week | 0
  Incidence of retrograde ejaculation at 1 Month | 0
  Incidence of retrograde ejaculation at 3 Months | 0

12. Secondary Outcome: International Prostate Symptom Score (IPSS) Assessment by Prostate Volume
Description: International Prostate Symptom Score (IPSS) scores were recorded at Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, then annually to 5 years. The mean change in IPSS was calculated. IPSS scores range from 0 (no symptoms) to 35 (severe symptoms). Mean change in IPSS scores reported at each follow-up interval. Improvement in symptoms is shown by a reduction in score.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Measure calculated for subjects providing data at each follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rezum Treatment - Larger Prostates (≥35gm); Rezum Treatment - Smaller Prostates (<35g): Subjects received the Rezum transurethral needle ablation procedure to treat benign prostatic hyperplasia.
  Rezum System: The Rezūm System treats patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death. The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
Arm/Group | Rezum Treatment - Larger Prostates (≥35gm) | Rezum Treatment - Smaller Prostates (<35g)
Number analyzed (Participants) | 37 | 13
score on a scale
  IPSS Change at 1 Week: number analyzed (Participants) | 36 | 13
  IPSS Change at 1 Week | 0.3 (7.2) | -2.4 (9.3)
  IPSS Change at 1 Month: number analyzed (Participants) | 36 | 13
  IPSS Change at 1 Month | -3.4 (8.0) | -9.4 (7.8)
  IPSS Change at 3 Months: number analyzed (Participants) | 35 | 13
  IPSS Change at 3 Months | -12.0 (6.6) | -15.9 (8.3)
  IPSS Change at 6 Months: number analyzed (Participants) | 35 | 13
  IPSS Change at 6 Months | -11.8 (7.1) | -14.9 (9.7)
  IPSS Change at 12 Months: number analyzed (Participants) | 32 | 13
  IPSS Change at 12 Months | -11.6 (7.7) | -13.7 (8.0)
  IPSS Change at 24 Months: number analyzed (Participants) | 26 | 9
  IPSS Change at 24 Months | -10.2 (8.4) | -16.1 (7.4)
  IPSS Change at 36 Months: number analyzed (Participants) | 20 | 7
  IPSS Change at 36 Months | -9.2 (9.3) | 10.0 (8.8)
  IPSS Change at 48 Months: number analyzed (Participants) | 20 | 6
  IPSS Change at 48 Months | -9.6 (8.4) | -9.5 (4.0)
  IPSS Change at 60 Months: number analyzed (Participants) | 5 | 2
  IPSS Change at 60 Months | -6.0 (5.6) | -14.5 (6.4)

13. Secondary Outcome: International Prostate Symptom Score (IPSS) Assessment Based on Prostate Lobe Treated: Lateral Only vs. Lateral and Median Lobe
Description: International Prostate Symptom Score (IPSS) scores were recorded at Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, then annually to 5 years. The mean change in IPSS was calculated. IPSS scores range from 0 (no symptoms) to 35 (severe symptoms). Mean change in IPSS scores reported at each follow-up interval. Improvement in symptoms is shown by a reduction in score.
  Results report change in IPSS by follow up interval for subjects treated in both lateral lobes and median lobe vs. subjects treated in lateral lobes alone.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rezum Treatment - No Median Lobe Present (Lateral Lobes Treated); Rezum Treatment - Median Lobe Present (Lateral and Median Lobes Treated): Subjects received the Rezum transurethral needle ablation procedure to treat benign prostatic hyperplasia.
  Rezum System: The Rezūm System treats patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death. The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
Arm/Group | Rezum Treatment - No Median Lobe Present (Lateral Lobes Treated) | Rezum Treatment - Median Lobe Present (Lateral and Median Lobes Treated)
Number analyzed (Participants) | 37 | 13
score on a scale
  IPSS Change at 1 Week: number analyzed (Participants) | 36 | 13
  IPSS Change at 1 Week | 0.4 (7.6) | -2.5 (8.2)
  IPSS Change at 1 Month: number analyzed (Participants) | 36 | 13
  IPSS Change at 1 Month | -4.1 (7.0) | -7.4 (11.2)
  IPSS Change at 3 Months: number analyzed (Participants) | 37 | 11
  IPSS Change at 3 Months | -11.9 (6.7) | -17.0 (7.8)
  IPSS Change at 6 Months: number analyzed (Participants) | 37 | 11
  IPSS Change at 6 Months | -12.2 (7.5) | -14.3 (9.2)
  IPSS Change at 12 Months: number analyzed (Participants) | 34 | 11
  IPSS Change at 12 Months | -11.9 (7.5) | -13.1 (8.7)
  IPSS Change at 24 Months: number analyzed (Participants) | 26 | 9
  IPSS Change at 24 Months | 11.7 (7.7) | -11.8 (10.9)
  IPSS Change at 36 Months: number analyzed (Participants) | 21 | 6
  IPSS Change at 36 Months | -9.4 (8.9) | -9.2 (10.2)
  IPSS Change at 48 Months: number analyzed (Participants) | 21 | 5
  IPSS Change at 48 Months | -10.5 (7.4) | -5.6 (7.5)
  IPSS Change at 60 Months: number analyzed (Participants) | 6 | 1
  IPSS Change at 60 Months | -8.2 (7.3) | -10.0 (0.0)

14. Secondary Outcome: International Prostate Symptom Score (IPSS) Assessment Based on Baseline IPSS
Description: International Prostate Symptom Score (IPSS) scores were recorded at Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, then annually to 5 years. The mean change in IPSS was calculated. IPSS scores range from 0 (no symptoms) to 35 (severe symptoms). Mean change in IPSS scores reported at each follow-up interval and grouped by Baseline IPSS. Improvement in symptoms is shown by a reduction in score.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Subjects With Baseline IPSS 13-19; Subjects With Baseline IPSS 20-25; Subjects With Baseline IPSS 26-35: Subjects received the Rezum transurethral needle ablation procedure to treat benign prostatic hyperplasia.
  Rezum System: The Rezūm System treats patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death. The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
Arm/Group | Subjects With Baseline IPSS 13-19 | Subjects With Baseline IPSS 20-25 | Subjects With Baseline IPSS 26-35
Number analyzed (Participants) | 23 | 20 | 7
score on a scale
  IPSS Change at 1 Week: number analyzed (Participants) | 22 | 20 | 7
  IPSS Change at 1 Week | 1.8 (4.9) | -2.9 (9.1) | -0.1 (10.2)
  IPSS Change at 1 Month: number analyzed (Participants) | 22 | 20 | 7
  IPSS Change at 1 Month | -3.3 (7.0) | -5.4 (8.7) | -9.0 (10.6)
  IPSS Change at 3 Months: number analyzed (Participants) | 22 | 19 | 7
  IPSS Change at 3 Months | -9.7 (5.4) | -13.9 (7.1) | -21.4 (5.5)
  IPSS Change at 6 Months: number analyzed (Participants) | 22 | 19 | 7
  IPSS Change at 6 Months | -9.2 (5.8) | -14.1 (7.7) | -19.7 (8.9)
  IPSS Change at 12 Months: number analyzed (Participants) | 21 | 18 | 6
  IPSS Change at 12 Months | -8.2 (5.0) | -14.6 (7.6) | -19.2 (9.2)
  IPSS Change at 24 Months: number analyzed (Participants) | 16 | 14 | 5
  IPSS Change at 24 Months | -7.9 (5.2) | -12.9 (8.9) | -20.6 (9.2)
  IPSS Change at 36 Months: number analyzed (Participants) | 12 | 12 | 3
  IPSS Change at 36 Months | -6.9 (5.2) | -9.0 (10.9) | -20.7 (4.0)
  IPSS Change at 48 Months: number analyzed (Participants) | 11 | 12 | 3
  IPSS Change at 48 Months | -7.2 (5.2) | -9.8 (8.3) | -17.7 (8.0)
  IPSS Change at 60 Months: number analyzed (Participants) | 3 | 2 | 2
  IPSS Change at 60 Months | -7.7 (4.7) | -3.5 (7.8) | -14.5 (6.4)

15. Secondary Outcome: Procedural Pain Score
Description: Pain scores were obtained for all subjects using the Iowa Pain Thermometer. Maximum intraprocedural pain scores were analyzed, together with the pain scores reported at follow-up intervals through 3 months. The treatment pain scores were reported by subjects post-procedure and was based on their recollections. Scale is 0-12 with higher scores corresponding to higher pain reported.
Time Frame: Day of treatment, 1 Day post procedure, 1 Week post procedure, 1 Month post procedure, 3 Months post procedure
Population: Subjects with data at the scheduled visits are included in the data summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  Pain Score on day of Treatment: number analyzed (Participants) | 45
  Pain Score on day of Treatment | 4.0 (3.3)
  Pain Score 1 Day Post-Treatment | 1.9 (2.3)
  Pain Score 1 Week Post-Treatment: number analyzed (Participants) | 48
  Pain Score 1 Week Post-Treatment | 1.9 (2.6)
  Pain Score 1 Month Post-Treatment: number analyzed (Participants) | 48
  Pain Score 1 Month Post-Treatment | 1.2 (2.1)
  Pain Score 3 Months Post-Treatment: number analyzed (Participants) | 43
  Pain Score 3 Months Post-Treatment | 0.5 (1.6)

16. Secondary Outcome: Quality of Life (QoL) - Change in QoL as Measured With the International Prostate Symptom Score (IPSS)
Description: Change in Quality of Life was measured using a QoL question in the IPSS. QoL data were collected at each follow up visit.
  One question in the IPSS asked subjects to rate their "quality of life due to urinary symptoms" on a scale of 0 = Delighted to 6 = Terrible.
  A reduction in score from baseline equates to improved outcome.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, then annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  Change from Baseline in IPSS QoL Score at 1 Week: number analyzed (Participants) | 49
  Change from Baseline in IPSS QoL Score at 1 Week | -0.3 (1.4)
  Change from Baseline in IPSS QoL Score at 1 Month: number analyzed (Participants) | 49
  Change from Baseline in IPSS QoL Score at 1 Month | -1.1 (1.8)
  Change from Baseline in IPSS QoL Score at 3 Months: number analyzed (Participants) | 48
  Change from Baseline in IPSS QoL Score at 3 Months | -2.7 (1.6)
  Change from Baseline in IPSS QoL Score at 6 Months: number analyzed (Participants) | 48
  Change from Baseline in IPSS QoL Score at 6 Months | -2.7 (1.7)
  Change from Baseline in IPSS QoL Score at 12 Months: number analyzed (Participants) | 45
  Change from Baseline in IPSS QoL Score at 12 Months | -2.7 (1.5)
  Change in IPSS QoL Change from Baseline in IPSS QoL Score at 24 Months: number analyzed (Participants) | 35
  Change in IPSS QoL Change from Baseline in IPSS QoL Score at 24 Months | -2.6 (1.7)
  Change from Baseline in IPSS QoL Score at 36 Months: number analyzed (Participants) | 27
  Change from Baseline in IPSS QoL Score at 36 Months | -2.4 (2.1)
  Change from Baseline in IPSS QoL Score at 48 Months: number analyzed (Participants) | 26
  Change from Baseline in IPSS QoL Score at 48 Months | -2.5 (1.6)
  Change from Baseline in IPSS QoL Score at 60 Months: number analyzed (Participants) | 7
  Change from Baseline in IPSS QoL Score at 60 Months | -1.6 (1.8)

17. Secondary Outcome: Quality of Life (QoL) - Change in QoL as Measured With the Benign Prostatic Hyperplasia Impact Index (BPHII)
Description: Change in Quality of Life will be measured with the Benign Prostatic Hyperplasia Impact Index (BPHII). Data were collected at specified follow up visits.
  BPHII scores range from 0 (no/mild symptoms) to 35 (severe symptoms). A reduction in score from baseline equates to an improvement in symptoms.
Time Frame: Baseline to 1 month, 3 months, 6 months, 1 year, then annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  Change from Baseline in BPHII Score at 1 Month: number analyzed (Participants) | 47
  Change from Baseline in BPHII Score at 1 Month | -1.0 (3.7)
  Change from Baseline in BPHII Score at 3 Months: number analyzed (Participants) | 47
  Change from Baseline in BPHII Score at 3 Months | -4.4 (2.9)
  Change from Baseline in BPHII Score at 6 Months: number analyzed (Participants) | 45
  Change from Baseline in BPHII Score at 6 Months | -4.5 (3.1)
  Change from Baseline in BPHII Score at 12 Months: number analyzed (Participants) | 43
  Change from Baseline in BPHII Score at 12 Months | -4.3 (2.8)
  Change from Baseline in BPHII Score at 24 Months: number analyzed (Participants) | 34
  Change from Baseline in BPHII Score at 24 Months | -4.4 (3.2)
  Change from Baseline in BPHII Score at 36 Months: number analyzed (Participants) | 26
  Change from Baseline in BPHII Score at 36 Months | -3.5 (4.0)
  Change from Baseline in BPHII Score at 48 Months: number analyzed (Participants) | 25
  Change from Baseline in BPHII Score at 48 Months | -4.0 (3.5)
  Change from Baseline in BPHII Score at 60 Months: number analyzed (Participants) | 7
  Change from Baseline in BPHII Score at 60 Months | -2.1 (4.2)

18. Secondary Outcome: Quality of Life (QoL) - Change in QoL as Measured With the EQ-5D-3L
Description: Quality of Life was measured using EQ-5D-3L questionnaire. QoL data were collected at each follow up visit. The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to all subjects to assess the effect of the treatment on the subjects' quality of life. EQ-5D-3L index ranges from -0.109 to 1.000, with 1.000 corresponding to the best health state and -0.109 corresponding to the worst health. Mean change in overall score from baseline is reported.
Time Frame: 1 month, 3 months, 6 months, 1 year, then annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  Change from Baseline in EQ-5D-3L Overall Score at 1 Month: number analyzed (Participants) | 47
  Change from Baseline in EQ-5D-3L Overall Score at 1 Month | -0.0 (0.2)
  Change from Baseline in EQ-5D-3L Overall Score at 3 Month: number analyzed (Participants) | 47
  Change from Baseline in EQ-5D-3L Overall Score at 3 Month | 0.0 (0.2)
  Change from Baseline in EQ-5D-3L Overall Score at 6 Month: number analyzed (Participants) | 46
  Change from Baseline in EQ-5D-3L Overall Score at 6 Month | 0.1 (0.1)
  Change from Baseline in EQ-5D-3L Overall Score at 12 Month: number analyzed (Participants) | 44
  Change from Baseline in EQ-5D-3L Overall Score at 12 Month | 0.0 (0.1)
  Change from Baseline in EQ-5D-3L Overall Score at 24 Month: number analyzed (Participants) | 33
  Change from Baseline in EQ-5D-3L Overall Score at 24 Month | 0.0 (0.1)
  Change from Baseline in EQ-5D-3L Overall Score at 36 Month: number analyzed (Participants) | 27
  Change from Baseline in EQ-5D-3L Overall Score at 36 Month | 0.0 (0.1)
  Change from Baseline in EQ-5D-3L Overall Score at 48 Month: number analyzed (Participants) | 26
  Change from Baseline in EQ-5D-3L Overall Score at 48 Month | -0.0 (0.2)
  Change from Baseline in EQ-5D-3L Overall Score at 60 Month: number analyzed (Participants) | 7
  Change from Baseline in EQ-5D-3L Overall Score at 60 Month | -0.1 (0.1)

19. Secondary Outcome: Quality of Life (QoL) - Change in QoL as Measured With the EQ-5D-3L Visual Analog Scale (VAS)
Description: Quality of Life was measured using EQ-5D-3L questionnaire and collected at each follow up visit. The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to all subjects to assess the effect of the treatment on the subjects' quality of life. The EQ-5D-3L includes a visual analog scale (VAS) which is a vertical scale with numbers ranging from 0 to 100. Subjects were asked to draw a line to the place on the scale that best represented how good or bad his health was on that day. The worst state a subject can imagine is marked zero, and the best state the subject can imagine is marked 100. Mean change in VAS score from baseline is reported. An increase in score is considered a better outcome.
Time Frame: 1 month, 3 months, 6 months, 1 year, then annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
score on a scale
  Change from Baseline in EQ-5D-3L VAS Score at 1 Month: number analyzed (Participants) | 42
  Change from Baseline in EQ-5D-3L VAS Score at 1 Month | 2.8 (18.0)
  Change from Baseline in EQ-5D-3L VAS Score at 3 Month: number analyzed (Participants) | 47
  Change from Baseline in EQ-5D-3L VAS Score at 3 Month | 8.3 (18.3)
  Change from Baseline in EQ-5D-3L VAS Score at 6 Month: number analyzed (Participants) | 47
  Change from Baseline in EQ-5D-3L VAS Score at 6 Month | 9.1 (14.5)
  Change from Baseline in EQ-5D-3L VAS Score at 12 Month: number analyzed (Participants) | 45
  Change from Baseline in EQ-5D-3L VAS Score at 12 Month | 7.4 (19.7)
  Change from Baseline in EQ-5D-3L VAS Score at 24 Month: number analyzed (Participants) | 34
  Change from Baseline in EQ-5D-3L VAS Score at 24 Month | 5.8 (18.3)
  Change from Baseline in EQ-5D-3L VAS Score at 36 Month: number analyzed (Participants) | 27
  Change from Baseline in EQ-5D-3L VAS Score at 36 Month | 9.2 (20.9)
  -0.1Change from Baseline in EQ-5D-3L VAS Score at 48 Month: number analyzed (Participants) | 26
  -0.1Change from Baseline in EQ-5D-3L VAS Score at 48 Month | 6.5 (17.9)
  Change from Baseline in EQ-5D-3L VAS Score at 60 Month: number analyzed (Participants) | 7
  Change from Baseline in EQ-5D-3L VAS Score at 60 Month | -0.1 (11.9)

20. Secondary Outcome: Quality of Life (QoL) - QoL Dimensions as Measured With the EQ-5D-3L
Description: Quality of Life was measured using EQ-5D-3L questionnaire. QoL data were collected at each follow up visit. The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to all subjects to assess the effect of the treatment on the subjects' quality of life. Each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =severe problems) in the relevant health dimension.
  Presented below are the scoring counts for each of the dimensions for baseline and follow up interval.
Time Frame: 1 month, 3 months, 6 months, 1 year, then annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Baseline_Anxiety Dimension Score: Level 1 (No Problems) | 32
  Baseline_Anxiety Dimension Score: Level 2 (Some Problems) | 16
  Baseline_Anxiety Dimension Score: Level 3 (Extreme Problems) | 2
  1 Month_Anxiety Dimension Score: number analyzed (Participants) | 49
  1 Month_Anxiety Dimension Score: Level 1 (No Problems) | 39
  1 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 8
  1 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 2
  3 Month_Anxiety Dimension Score: number analyzed (Participants) | 47
  3 Month_Anxiety Dimension Score: Level 1 (No Problems) | 41
  3 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 6
  3 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  6 Month_Anxiety Dimension Score: number analyzed (Participants) | 46
  6 Month_Anxiety Dimension Score: Level 1 (No Problems) | 40
  6 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 6
  6 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  12 Month_Anxiety Dimension Score: number analyzed (Participants) | 45
  12 Month_Anxiety Dimension Score: Level 1 (No Problems) | 35
  12 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 10
  12 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  24 Month_Anxiety Dimension Score: number analyzed (Participants) | 34
  24 Month_Anxiety Dimension Score: Level 1 (No Problems) | 26
  24 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 8
  24 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  36 Month_Anxiety Dimension Score: number analyzed (Participants) | 27
  36 Month_Anxiety Dimension Score: Level 1 (No Problems) | 22
  36 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 5
  36 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  48 Month_Anxiety Dimension Score: number analyzed (Participants) | 26
  48 Month_Anxiety Dimension Score: Level 1 (No Problems) | 19
  48 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 7
  48 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  60 Month_Anxiety Dimension Score: number analyzed (Participants) | 7
  60 Month_Anxiety Dimension Score: Level 1 (No Problems) | 5
  60 Month_Anxiety Dimension Score: Level 2 (Some Problems) | 2
  60 Month_Anxiety Dimension Score: Level 3 (Extreme Problems) | 0
  Baseline_Mobility Dimension Score: Level 1 (No Problems) | 43
  Baseline_Mobility Dimension Score: Level 2 (Some Problems) | 7
  Baseline_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  1 Month_Mobility Dimension Score: number analyzed (Participants) | 49
  1 Month_Mobility Dimension Score: Level 1 (No Problems) | 43
  1 Month_Mobility Dimension Score: Level 2 (Some Problems) | 6
  1 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  3 Month_Mobility Dimension Score: number analyzed (Participants) | 48
  3 Month_Mobility Dimension Score: Level 1 (No Problems) | 43
  3 Month_Mobility Dimension Score: Level 2 (Some Problems) | 5
  3 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  6 Month_Mobility Dimension Score: number analyzed (Participants) | 46
  6 Month_Mobility Dimension Score: Level 1 (No Problems) | 40
  6 Month_Mobility Dimension Score: Level 2 (Some Problems) | 6
  6 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  12 Month_Mobility Dimension Score: number analyzed (Participants) | 45
  12 Month_Mobility Dimension Score: Level 1 (No Problems) | 37
  12 Month_Mobility Dimension Score: Level 2 (Some Problems) | 8
  12 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  24 Month_Mobility Dimension Score: number analyzed (Participants) | 34
  24 Month_Mobility Dimension Score: Level 1 (No Problems) | 27
  24 Month_Mobility Dimension Score: Level 2 (Some Problems) | 7
  24 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  36 Month_Mobility Dimension Score: number analyzed (Participants) | 27
  36 Month_Mobility Dimension Score: Level 1 (No Problems) | 17
  36 Month_Mobility Dimension Score: Level 2 (Some Problems) | 10
  36 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  48 Month_Mobility Dimension Score: number analyzed (Participants) | 25
  48 Month_Mobility Dimension Score: Level 1 (No Problems) | 15
  48 Month_Mobility Dimension Score: Level 2 (Some Problems) | 10
  48 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  60 Month_Mobility Dimension Score: number analyzed (Participants) | 7
  60 Month_Mobility Dimension Score: Level 1 (No Problems) | 3
  60 Month_Mobility Dimension Score: Level 2 (Some Problems) | 4
  60 Month_Mobility Dimension Score: Level 3 (Extreme Problems) | 0
  Baseline_Pain Dimension Score: number analyzed (Participants) | 48
  Baseline_Pain Dimension Score: Level 1 (No Problems) | 22
  Baseline_Pain Dimension Score: Level 2 (Some Problems) | 25
  Baseline_Pain Dimension Score: Level 3 (Extreme Problems) | 1
  1 Month_Pain Dimension Score: number analyzed (Participants) | 46
  1 Month_Pain Dimension Score: Level 1 (No Problems) | 24
  1 Month_Pain Dimension Score: Level 2 (Some Problems) | 20
  1 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 2
  3 Month_Pain Dimension Score: number analyzed (Participants) | 48
  3 Month_Pain Dimension Score: Level 1 (No Problems) | 32
  3 Month_Pain Dimension Score: Level 2 (Some Problems) | 15
  3 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 1
  6 Month_Pain Dimension Score: number analyzed (Participants) | 46
  6 Month_Pain Dimension Score: Level 1 (No Problems) | 30
  6 Month_Pain Dimension Score: Level 2 (Some Problems) | 16
  6 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 0
  12 Month_Pain Dimension Score: number analyzed (Participants) | 44
  12 Month_Pain Dimension Score: Level 1 (No Problems) | 28
  12 Month_Pain Dimension Score: Level 2 (Some Problems) | 16
  12 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 0
  24 Month_Pain Dimension Score: number analyzed (Participants) | 33
  24 Month_Pain Dimension Score: Level 1 (No Problems) | 20
  24 Month_Pain Dimension Score: Level 2 (Some Problems) | 12
  24 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 1
  36 Month_Pain Dimension Score: number analyzed (Participants) | 27
  36 Month_Pain Dimension Score: Level 1 (No Problems) | 17
  36 Month_Pain Dimension Score: Level 2 (Some Problems) | 9
  36 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 1
  48 Month_Pain Dimension Score: number analyzed (Participants) | 26
  48 Month_Pain Dimension Score: Level 1 (No Problems) | 12
  48 Month_Pain Dimension Score: Level 2 (Some Problems) | 12
  48 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 2
  60 Month_Pain Dimension Score: number analyzed (Participants) | 7
  60 Month_Pain Dimension Score: Level 1 (No Problems) | 4
  60 Month_Pain Dimension Score: Level 2 (Some Problems) | 2
  60 Month_Pain Dimension Score: Level 3 (Extreme Problems) | 1
  Baseline_Self-care Dimension Score: Level 1 (No Problems) | 50
  Baseline_Self-care Dimension Score: Level 2 (Some Problems) | 0
  Baseline_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  1 Month_Self-care Dimension Score: number analyzed (Participants) | 49
  1 Month_Self-care Dimension Score: Level 1 (No Problems) | 48
  1 Month_Self-care Dimension Score: Level 2 (Some Problems) | 0
  1 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 1
  3 Month_Self-care Dimension Score: number analyzed (Participants) | 48
  3 Month_Self-care Dimension Score: Level 1 (No Problems) | 47
  3 Month_Self-care Dimension Score: Level 2 (Some Problems) | 1
  3 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  6 Month_Self-care Dimension Score: number analyzed (Participants) | 46
  6 Month_Self-care Dimension Score: Level 1 (No Problems) | 46
  6 Month_Self-care Dimension Score: Level 2 (Some Problems) | 0
  6 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  12 Month_Self-care Dimension Score: number analyzed (Participants) | 45
  12 Month_Self-care Dimension Score: Level 1 (No Problems) | 45
  12 Month_Self-care Dimension Score: Level 2 (Some Problems) | 0
  12 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  24 Month_Self-care Dimension Score: number analyzed (Participants) | 34
  24 Month_Self-care Dimension Score: Level 1 (No Problems) | 33
  24 Month_Self-care Dimension Score: Level 2 (Some Problems) | 1
  24 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  36 Month_Self-care Dimension Score: number analyzed (Participants) | 27
  36 Month_Self-care Dimension Score: Level 1 (No Problems) | 26
  36 Month_Self-care Dimension Score: Level 2 (Some Problems) | 1
  36 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  48 Month_Self-care Dimension Score: number analyzed (Participants) | 25
  48 Month_Self-care Dimension Score: Level 1 (No Problems) | 24
  48 Month_Self-care Dimension Score: Level 2 (Some Problems) | 1
  48 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  60 Month_Self-care Dimension Score: number analyzed (Participants) | 7
  60 Month_Self-care Dimension Score: Level 1 (No Problems) | 6
  60 Month_Self-care Dimension Score: Level 2 (Some Problems) | 1
  60 Month_Self-care Dimension Score: Level 3 (Extreme Problems) | 0
  Baseline_Usual Activity Dimension Score: Level 1 (No Problems) | 47
  Baseline_Usual Activity Dimension Score: Level 2 (Some Problems) | 3
  Baseline_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0
  1 Month_Usual Activity Dimension Score: number analyzed (Participants) | 49
  1 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 40
  1 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 7
  1 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 2
  3 Month_Usual Activity Dimension Score: number analyzed (Participants) | 48
  3 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 45
  3 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 3
  3 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0
  6 Month_Usual Activity Dimension Score: number analyzed (Participants) | 46
  6 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 46
  6 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 0
  6 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0
  12 Month_Usual Activity Dimension Score: number analyzed (Participants) | 45
  12 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 41
  12 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 4
  12 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0
  24 Month_Usual Activity Dimension Score: number analyzed (Participants) | 34
  24 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 31
  24 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 3
  24 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0
  36 Month_Usual Activity Dimension Score: number analyzed (Participants) | 27
  36 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 25
  36 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 2
  36 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0
  48 Month_Usual Activity Dimension Score: number analyzed (Participants) | 25
  48 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 20
  48 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 4
  48 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 1
  60 Month_Usual Activity Dimension Score: number analyzed (Participants) | 7
  60 Month_Usual Activity Dimension Score: Level 1 (No Problems) | 6
  60 Month_Usual Activity Dimension Score: Level 2 (Some Problems) | 1
  60 Month_Usual Activity Dimension Score: Level 3 (Extreme Problems) | 0

21. Secondary Outcome: Subject Satisfaction - Satisfied With Overall Procedure
Description: Subject satisfaction assessed using a study specific questionnaire to evaluate the subject's overall satisfaction of the procedure at 1 week, 1 month, 3 months, 6 months, 1 year, and annually to 5 years.
  These will be measured as:
  • Proportion of subjects that are satisfied with the procedure overall
  Note: Subject Satisfaction Questionnaire is specific to the NxThera Rezūm treatment and 3 of the 7 questions were used to evaluate the subjects' overall satisfaction with the procedure. Within the questionnaire, subjects sometimes did not answer all of the questions, which resulted in a different "n" by question within the same follow-up time point.
Time Frame: 1 week, 1 month, 3 months, 6 months, 1 year, and annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Proportion of subjects satisfied with the procedure at 1 Week: number analyzed (Participants) | 48
  Proportion of subjects satisfied with the procedure at 1 Week: Very Satisfied | 16
  Proportion of subjects satisfied with the procedure at 1 Week: Satisfied | 23
  Proportion of subjects satisfied with the procedure at 1 Week: Neither Satisfied or Dissatisfied (Neutral) | 6
  Proportion of subjects satisfied with the procedure at 1 Week: Dissatisfied | 2
  Proportion of subjects satisfied with the procedure at 1 Week: Very Dissatisfied | 1
  Proportion of subjects satisfied with the procedure at 1 Month: number analyzed (Participants) | 47
  Proportion of subjects satisfied with the procedure at 1 Month: Very Satisfied | 18
  Proportion of subjects satisfied with the procedure at 1 Month: Satisfied | 19
  Proportion of subjects satisfied with the procedure at 1 Month: Neither Satisfied or Dissatisfied (Neutral) | 8
  Proportion of subjects satisfied with the procedure at 1 Month: Dissatisfied | 2
  Proportion of subjects satisfied with the procedure at 1 Month: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 3 Months: number analyzed (Participants) | 47
  Proportion of subjects satisfied with the procedure at 3 Months: Very Satisfied | 21
  Proportion of subjects satisfied with the procedure at 3 Months: Satisfied | 22
  Proportion of subjects satisfied with the procedure at 3 Months: Neither Satisfied or Dissatisfied (Neutral) | 3
  Proportion of subjects satisfied with the procedure at 3 Months: Dissatisfied | 1
  Proportion of subjects satisfied with the procedure at 3 Months: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 6 Months: number analyzed (Participants) | 47
  Proportion of subjects satisfied with the procedure at 6 Months: Very Satisfied | 18
  Proportion of subjects satisfied with the procedure at 6 Months: Satisfied | 20
  Proportion of subjects satisfied with the procedure at 6 Months: Neither Satisfied or Dissatisfied (Neutral) | 7
  Proportion of subjects satisfied with the procedure at 6 Months: Dissatisfied | 2
  Proportion of subjects satisfied with the procedure at 6 Months: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 12 Months: number analyzed (Participants) | 45
  Proportion of subjects satisfied with the procedure at 12 Months: Very Satisfied | 19
  Proportion of subjects satisfied with the procedure at 12 Months: Satisfied | 19
  Proportion of subjects satisfied with the procedure at 12 Months: Neither Satisfied or Dissatisfied (Neutral) | 6
  Proportion of subjects satisfied with the procedure at 12 Months: Dissatisfied | 1
  Proportion of subjects satisfied with the procedure at 12 Months: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 24 Months: number analyzed (Participants) | 27
  Proportion of subjects satisfied with the procedure at 24 Months: Very Satisfied | 12
  Proportion of subjects satisfied with the procedure at 24 Months: Satisfied | 12
  Proportion of subjects satisfied with the procedure at 24 Months: Neither Satisfied or Dissatisfied (Neutral) | 3
  Proportion of subjects satisfied with the procedure at 24 Months: Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 24 Months: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 36 Months: number analyzed (Participants) | 23
  Proportion of subjects satisfied with the procedure at 36 Months: Very Satisfied | 11
  Proportion of subjects satisfied with the procedure at 36 Months: Satisfied | 8
  Proportion of subjects satisfied with the procedure at 36 Months: Neither Satisfied or Dissatisfied (Neutral) | 4
  Proportion of subjects satisfied with the procedure at 36 Months: Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 36 Months: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 48 Months: number analyzed (Participants) | 26
  Proportion of subjects satisfied with the procedure at 48 Months: Very Satisfied | 10
  Proportion of subjects satisfied with the procedure at 48 Months: Satisfied | 11
  Proportion of subjects satisfied with the procedure at 48 Months: Neither Satisfied or Dissatisfied (Neutral) | 3
  Proportion of subjects satisfied with the procedure at 48 Months: Dissatisfied | 2
  Proportion of subjects satisfied with the procedure at 48 Months: Very Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 60 Months: number analyzed (Participants) | 7
  Proportion of subjects satisfied with the procedure at 60 Months: Very Satisfied | 1
  Proportion of subjects satisfied with the procedure at 60 Months: Satisfied | 4
  Proportion of subjects satisfied with the procedure at 60 Months: Neither Satisfied or Dissatisfied (Neutral) | 2
  Proportion of subjects satisfied with the procedure at 60 Months: Dissatisfied | 0
  Proportion of subjects satisfied with the procedure at 60 Months: Very Dissatisfied | 0

22. Secondary Outcome: Subject Satisfaction - Proportion of Subjects Who Would Recommend Procedure to Friends and Family
Description: Subject satisfaction assessed using a study specific questionnaire to evaluate the subject's overall satisfaction of the procedure at 1 week, 1 month, 3 months, 6 months, 1 year, and annually to 5 years.
  Outcome measured as:
  • Proportion of subjects that would recommend this treatment to friends and families
  Note: Subject Satisfaction Questionnaire is specific to the NxThera Rezūm treatment and 3 of the 7 questions were used to evaluate the subjects' overall satisfaction with the procedure. Within the questionnaire, subjects sometimes did not answer all of the questions, which resulted in a different "n" by question within the same follow-up time point.
Time Frame: 1 week, 1 month, 3 months, 6 months, 1 year, and annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Proportion of subjects who would recommend procedure to friends/family at 1 Week: number analyzed (Participants) | 48
  Proportion of subjects who would recommend procedure to friends/family at 1 Week: Definitely Will | 26
  Proportion of subjects who would recommend procedure to friends/family at 1 Week: Probably Will | 14
  Proportion of subjects who would recommend procedure to friends/family at 1 Week: Not Sure | 7
  Proportion of subjects who would recommend procedure to friends/family at 1 Week: Probably Will Not | 1
  Proportion of subjects who would recommend procedure to friends/family at 1 Week: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 1 Month: number analyzed (Participants) | 48
  Proportion of subjects who would recommend procedure to friends/family at 1 Month: Definitely Will | 24
  Proportion of subjects who would recommend procedure to friends/family at 1 Month: Probably Will | 16
  Proportion of subjects who would recommend procedure to friends/family at 1 Month: Not Sure | 6
  Proportion of subjects who would recommend procedure to friends/family at 1 Month: Probably Will Not | 2
  Proportion of subjects who would recommend procedure to friends/family at 1 Month: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 3 Months: number analyzed (Participants) | 48
  Proportion of subjects who would recommend procedure to friends/family at 3 Months: Definitely Will | 33
  Proportion of subjects who would recommend procedure to friends/family at 3 Months: Probably Will | 10
  Proportion of subjects who would recommend procedure to friends/family at 3 Months: Not Sure | 4
  Proportion of subjects who would recommend procedure to friends/family at 3 Months: Probably Will Not | 1
  Proportion of subjects who would recommend procedure to friends/family at 3 Months: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 6 Months: number analyzed (Participants) | 47
  Proportion of subjects who would recommend procedure to friends/family at 6 Months: Definitely Will | 29
  Proportion of subjects who would recommend procedure to friends/family at 6 Months: Probably Will | 12
  Proportion of subjects who would recommend procedure to friends/family at 6 Months: Not Sure | 5
  Proportion of subjects who would recommend procedure to friends/family at 6 Months: Probably Will Not | 1
  Proportion of subjects who would recommend procedure to friends/family at 6 Months: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 12 Months: number analyzed (Participants) | 45
  Proportion of subjects who would recommend procedure to friends/family at 12 Months: Definitely Will | 30
  Proportion of subjects who would recommend procedure to friends/family at 12 Months: Probably Will | 12
  Proportion of subjects who would recommend procedure to friends/family at 12 Months: Not Sure | 3
  Proportion of subjects who would recommend procedure to friends/family at 12 Months: Probably Will Not | 0
  Proportion of subjects who would recommend procedure to friends/family at 12 Months: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 24 Months: number analyzed (Participants) | 27
  Proportion of subjects who would recommend procedure to friends/family at 24 Months: Definitely Will | 18
  Proportion of subjects who would recommend procedure to friends/family at 24 Months: Probably Will | 8
  Proportion of subjects who would recommend procedure to friends/family at 24 Months: Not Sure | 1
  Proportion of subjects who would recommend procedure to friends/family at 24 Months: Probably Will Not | 0
  Proportion of subjects who would recommend procedure to friends/family at 24 Months: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 36 Months: number analyzed (Participants) | 23
  Proportion of subjects who would recommend procedure to friends/family at 36 Months: Definitely Will | 17
  Proportion of subjects who would recommend procedure to friends/family at 36 Months: Probably Will | 5
  Proportion of subjects who would recommend procedure to friends/family at 36 Months: Not Sure | 1
  Proportion of subjects who would recommend procedure to friends/family at 36 Months: Probably Will Not | 0
  Proportion of subjects who would recommend procedure to friends/family at 36 Months: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 48 Months: number analyzed (Participants) | 26
  Proportion of subjects who would recommend procedure to friends/family at 48 Months: Definitely Will | 17
  Proportion of subjects who would recommend procedure to friends/family at 48 Months: Probably Will | 8
  Proportion of subjects who would recommend procedure to friends/family at 48 Months: Not Sure | 1
  Proportion of subjects who would recommend procedure to friends/family at 48 Months: Probably Will Not | 0
  Proportion of subjects who would recommend procedure to friends/family at 48 Months: Definitely Will not | 0
  Proportion of subjects who would recommend procedure to friends/family at 60 Months: number analyzed (Participants) | 7
  Proportion of subjects who would recommend procedure to friends/family at 60 Months: Definitely Will | 4
  Proportion of subjects who would recommend procedure to friends/family at 60 Months: Probably Will | 1
  Proportion of subjects who would recommend procedure to friends/family at 60 Months: Not Sure | 2
  Proportion of subjects who would recommend procedure to friends/family at 60 Months: Probably Will Not | 0
  Proportion of subjects who would recommend procedure to friends/family at 60 Months: Definitely Will not | 0

23. Secondary Outcome: Subject Satisfaction - Proportion of Subjects Who Would Undergo Same Treatment if Symptoms Were to Recur After 5 Years
Description: Subject satisfaction assessed using a study specific questionnaire to evaluate the subject's overall satisfaction of the procedure at 1 week, 1 month, 3 months, 6 months, 1 year, and annually to 5 years.
  Outcome measured as:
  • Proportion of subjects who would undergo the same treatment if their symptoms were to recur after 5 years
  Note: Subject Satisfaction Questionnaire is specific to the NxThera Rezūm treatment and 3 of the 7 questions were used to evaluate the subjects' overall satisfaction with the procedure. Within the questionnaire, subjects sometimes did not answer all of the questions, which resulted in a different "n" by question within the same follow-up time point.
Time Frame: 1 week, 1 month, 3 months, 6 months, 1 year, and annually to 5 years
Population: Subjects with data at baseline and follow-up visit are included in the summarization.
Measure: Count of Participants; unit: Participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
Participants
  Subjects at 1 Week willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 47
  Subjects at 1 Week willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 23
  Subjects at 1 Week willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 17
  Subjects at 1 Week willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 6
  Subjects at 1 Week willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 1
  Subjects at 1 Week willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0
  Subjects at 1 Month willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 48
  Subjects at 1 Month willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 17
  Subjects at 1 Month willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 21
  Subjects at 1 Month willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 8
  Subjects at 1 Month willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 2
  Subjects at 1 Month willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0
  Subjects at 3 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 47
  Subjects at 3 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 27
  Subjects at 3 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 15
  Subjects at 3 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 5
  Subjects at 3 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 0
  Subjects at 3 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0
  Subjects at 6 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 47
  Subjects at 6 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 25
  Subjects at 6 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 13
  Subjects at 6 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 8
  Subjects at 6 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 1
  Subjects at 6 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0
  Subjects at 12 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 45
  Subjects at 12 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 29
  Subjects at 12 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 10
  Subjects at 12 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 5
  Subjects at 12 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 0
  Subjects at 12 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 1
  Subjects at 24 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 27
  Subjects at 24 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 12
  Subjects at 24 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 12
  Subjects at 24 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 2
  Subjects at 24 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 0
  Subjects at 24 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 1
  Subjects at 36 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 23
  Subjects at 36 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 10
  Subjects at 36 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 8
  Subjects at 36 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 2
  Subjects at 36 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 3
  Subjects at 36 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0
  Subjects at 48 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 26
  Subjects at 48 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 12
  Subjects at 48 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 8
  Subjects at 48 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 5
  Subjects at 48 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 1
  Subjects at 48 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0
  Subjects at 60 Months willing to undergo re-treatment in 5 years if symptoms were to recur: number analyzed (Participants) | 7
  Subjects at 60 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Likely | 1
  Subjects at 60 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Likely | 3
  Subjects at 60 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Not Sure | 3
  Subjects at 60 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Unlikely | 0
  Subjects at 60 Months willing to undergo re-treatment in 5 years if symptoms were to recur: Very Unlikely | 0

24. Secondary Outcome: Procedural Parameters - Procedure Time
Description: Procedure time: Time from delivery device insertion to final delivery device withdrawal
Time Frame: Day of Procedure
Population: Subjects with procedure data are included in the summarization.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
minutes | 6.7 (5.8)

25. Secondary Outcome: Procedural Parameters - Treatment Time
Description: Treatment time: time from first vapor delivery to last vapor delivery
Time Frame: Day of Procedure
Population: Subjects with procedure data are included in the summarization.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 50
minutes | 4.5 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of index procedure through the 60 month follow-up assessment.
Arm/Group | Rezum Treatment
All-Cause Mortality (participants affected / at risk) | 2/50
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rezum Treatment (N=50)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject had preexisting Congestive Heart Failure which deteriorated into symptomatic pulmonary edema, subject was hospitalized and treated.
Cardiac Event (Cardiac disorders) | 1 (1) — Subject with medical history of Hypertension, arrhythmia and diabetes, experienced a myocardial infarction and was hospitalized. A percutaneous transluminal coronary angiogram was done and subject was discharged home.
Pain/Discomfort - Pelvic (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject reported pain and discomfort in his right hip, and was hospitalized for a surgical revision of right hip endoprothesis coxae due to pain, and restricted, limited motion. The event was resolved after the revision procedure.
Urinary Retention (Renal and urinary disorders) | 3 (5) — Due to worsening urinary retention subject underwent TURP.
Urinary Frequency (Renal and urinary disorders) | 1 (1) — At one month follow up catheter was removed and subject voided, but later that day had a re-catheterization due to to urinary retention. Subject underwent cystoscopy and a prostatic median lobe was identified. Subject then had a TURP procedure.
Weakness or Fatigue (Gastrointestinal disorders) | 1 (1) — The subject reported having fatigue, weakness and diarrhea, and was hospitalized. The subject was diagnosed with Salmonella enteritis and treated with antibiotics.
Diarrhea (Gastrointestinal disorders) | 1 (1) — The subject reported having fatigue, weakness and diarrhea, and was hospitalized. The subject was diagnosed with Salmonella enteritis and treated with antibiotics.
Cancer -Other (Renal and urinary disorders) | 1 (1) — The subject reported undergoing a routine preventive colonoscopy and a tumor of the hepatic flexure in the colon was detected. Subject had a right hemi colectomy performed.
Urinary Tract Infection-Proven (Renal and urinary disorders) | 1 (1) — Subject reported sudden onset of fever (40C) and voided grayish appearing material. Subject hospitalized and was diagnosed with urosepsis. Subject was treated with Ciprofloxacin and event resolved.
Poor Stream (Renal and urinary disorders) | 1 (1) — At one month follow up catheter was removed and subject voided, but later that day had a re-catheterization due to to urinary retention. Subject underwent cystoscopy and a prostatic median lobe was identified. Subject then had a TURP procedure.
Other (General disorders) | 2 (5) — 002-005: Pain/Discomfort-Pelvic; R hip prosthesis revision; Gonarthrosis-subject underwent planned implantation of left knee endoptrothesis. 002-008: L arm pain (surgical repair of joint); Death due to previously unreported metastatic cancer
Infection Other than UTI (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rezum Treatment (N=50)
Urinary Retention (Renal and urinary disorders) | 15 (18)
Urinary Urgency (Renal and urinary disorders) | 15 (16)
Dysuria (Renal and urinary disorders) | 10 (10)
Other (General disorders) | 4 (5)
Poor Stream (Renal and urinary disorders) | 8 (9)
UTI - Suspected (Renal and urinary disorders) | 9 (10)
Nocturia (Renal and urinary disorders) | 6 (7)
Pain/Discomfort (General disorders) | 7 (7)
Hematuria - Gross (Renal and urinary disorders) | 4 (6)
Urinary Incontinence - Urge (Renal and urinary disorders) | 3 (5)
Urinary Frequency (Renal and urinary disorders) | 2 (3)
Hesitancy (Renal and urinary disorders) | 3 (3)
Pain/Discomfort - Pelvic (General disorders) | 1 (2)
Urethral Secretion w/o Hematuria or Stones (Renal and urinary disorders) | 3 (3)
Pain/Discomfort with Scrotum (Renal and urinary disorders) | 2 (2)
Abdominal Bloating with Gas (Gastrointestinal disorders) | 1 (1)
Bladder Spasms (Renal and urinary disorders) | 1 (1)
Cancer - Prostate (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Epididymitis (Skin and subcutaneous tissue disorders) | 1 (1)
Injury - Other (General disorders) | 1 (1)
Pain/Discomfort - Back (General disorders) | 1 (1)
Pain/Discomfort - Perineum (General disorders) | 1 (1)
Prostatic Cyst De Novo (Renal and urinary disorders) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Terminal Dribbling (Renal and urinary disorders) | 1 (1)
Urinary Incontinence - Not Specified (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a pilot study conducted on a new therapy at a limited number of sites (3 total).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No